CLINICAL TRIAL: NCT00239109
Title: Ziprasidone Versus Olanzapine In The Treatment Of Schizophrenia: A Six Months, Double Blind Randomized, Parallel Group Study.
Brief Title: Ziprasidone Versus Olanzapine In The Treatment Of Schizophrenia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281064
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone; Olanzapine; Weights and Measures

INTERVENTIONS:
Drug: Ziprasidone
Drug: Olanzapine
Procedure: Scales
Procedure: measures of the body (Weight...)
Procedure: Serum analysis

SUMMARY:
* Various studies suggest that patients treated with Olanzapine can experience a substantial weight gain, while no changes have been observed in patients treated with Ziprasidone. Negative consequences on lipid and glucose profiles have also been observed in patients treated with Olanzapine. Most of the available data belong to short-term studies. However, for most clinical trials the primary variable was an efficacy variable, and included the weight assessment as a secondary variable; they also lack a systematic monitoring of some variables that can play a role in weight gain, as the level of exercise, appetite increase, etc. and we have considered of importance their inclusion in this protocol. Previous studies did not assess visceral fat using widely standardized parameters as the waist index, which at certain levels is considered an indicator of the cardiovascular risk, or leptine, highly correlated to the body fat storage. We would like to fit the recently published American Diabetes Association, American Psychiatric Association, American Association of Clinical Endocrinologists and North American Association for the Study of Obesity Antipsychotic, obesity and diabetes mellitus consensus.22
* Schizophrenic patients show a 4-fold probability to die as a consequence of cardiovascular problems compared to the normal population. The antipsychotic treatment can contribute to increase this risk favoring weight gain and the appearance of cardiovascular risk factors associated to obesity (blood hypertension, hyperlipidemia, type II Diabetes Mellitus). We intend to obtain a complete cardiovascular risk profile of patients, as well as its change during antipsychotic treatment, including primary cardiovascular risk factors in addition to the analysis of markers that have recently been linked to cardiovascular risk (as reactive protein C).
* The study will evaluate the risk of hyperglycemia, insulin resistance and Diabetes Mellitus, and will investigate the association between glucose homeostasis abnormalities and weight gain in the treated patients. Likewise, adiponectine, secreted from adipocytes and a possible link between obesity and insulin resistance will be determined; recent studies show an adiponectine decrease in humans with insulin resistance and obesity; furthermore, prospective studies have shown these changes could predict a higher risk of DM development.
* Changes have been introduced in the complete evaluation of the patient's metabolic and cardiovascular profiles with the advice, and under the coordination of endocrinologists after a complete review of the subject

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of schizophrenia using the DSM-IV-TR criteria
* Patient's clinical condition should justify treatment initiation with a new antipsychotic drug.

Exclusion Criteria:

* Patients at immediate risk of committing harm to self or others
* Concurrent treatment with antipsychotic agents after randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2003-04; Study Completion 2007-02

PRIMARY OUTCOMES:
To estimate and compare the effects of ziprasidone vs olanzapine on body weight in the treatment of patients with schizophrenia.

SECONDARY OUTCOMES:
PANSS total score; change from baseline CGI severity; change from baseline CGI - Improvement PANSS negative subscale score; change from baseline DSM IV axis V Patient preference scale (PPS) Heath Utility Index Mark III BMI , Qaist Index

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Spain (7):
  - Pfizer Investigational Site, Bilbao, Vizcaya
  - Pfizer Investigational Site, Badajoz
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Salamanca
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Zamora

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281064&StudyName=Ziprasidone+Versus+Olanzapine+In+The+Treatment+Of+Schizophrenia%2E